CLINICAL TRIAL: NCT00519935
Title: Adherence to IDDM Regimen in Urban Youth
Brief Title: Testing MST to Improve Adherence Among Youth With Chronic Poor Metabolic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor, Wayne State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK59067A (completed); R01DK059067 (NIH)
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Dependent Diabetes Mellitus; family therapy; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multisystemic Therapy (Experimental): In-home, intensive family therapy
  Interventions: Behavioral: Multisystemic Therapy
- Standard Medical Care (TAU) (No Intervention): Standard medical care is provided at Children's Hospital of Michigan consistent with the standards for the care of children with T1D outlined by the American Diabetes Association.

INTERVENTIONS:
Behavioral: Multisystemic Therapy — MST is an individualized approach that begins with a comprehensive, multi-informant assessment that allows for the development of treatment goals and interventions that are individually tailored for each family. Therapists draw upon a menu of evidenced-based interventions that include cognitive-behavioral therapy, parent training and behavioral family systems therapy.
  Other Names: MST
  Arms: Multisystemic Therapy

SUMMARY:
The protocol is a randomized clinical trial providing Multisystemic Therapy (MST), an intensive home-based family psychotherapy intervention, to a group of urban adolescents with poorly controlled Type 1 diabetes and their families.

DETAILED DESCRIPTION:
Substantial data exists to demonstrate that improving metabolic control in persons with Type 1 diabetes mellitus (T1DM) can delay the onset of diabetes complications and reverse some existing complications as well. Unfortunately, those adolescents with T1DM who are at highest risk for diabetes complications are often the most resistant to hospital based care and traditional education/ supportive interventions. They are also faced with multiple barriers to improved metabolic control, which may include lack of knowledge about diabetes, family disorganization and disengagement, high levels of stress and an unhealthy lifestyle. Multisystemic Therapy (MST), a flexible and home-based therapeutic intervention originally designed for use with mental health populations, seems to be a promising approach to providing diabetic adolescents with the ability to engage in consistent and attentive illness management.

The study recruited a sample of 127 adolescents in poor metabolic control and randomly assigned them to either the treatment intervention, MST plus standard medical care, or standard medical care alone. Families randomized to MST received intensive, home-based family therapy for approximately six months. Families completed data collection at baseline and then again at 7, 12 18 and 24 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* a current hemoglobin A1c(HbA1c) of >8.0%
* an average HbA1c of >8.0% during the past year
* diagnosed with Type 1 diabetes for at least one year
* reside in the metro Detroit tri-county area

Exclusion Criteria:

* severe mental impairment/thought disorder
* non-English speaking patient/parent
* co-morbid major medical condition such as cystic fibrosis

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2001-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Control: Hemoglobin A1c (HbA1c) | 2 years
  Retrospective measure of blood glucose control, encompasses the previous 2-3 months

SECONDARY OUTCOMES:
Regimen Adherence: Diabetes Management Scale (DMS), Glucose Meter Downloads | 2 years
  The DMS assesses a broad range of management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision. Glucose meters only assess blood glucose monitoring, but are empirically linked to metabolic control.
DKA admissions and emergency room (ER) Visits: hospital information systems data extraction, Service Utilization Questionnaire (SUQ) | 2 years
  The number of patient visits to acute care settings represents a significant health care cost in this high-risk population.
Quality of life | 2 years
  44 scale item designed to tap life satisfaction, diabetes impact and diabetes related worries in adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Ellis, Ph.D., Principal Investigator — Wayne State University; Sylvie Naar-King, Ph.D., Principal Investigator — Wayne State University; Maureen O. Frey, Ph.D., Principal Investigator — Children's Hospital of Michigan
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ellis DA, Frey MA, Naar-King S, Templin T, Cunningham P, Cakan N. Use of multisystemic therapy to improve regimen adherence among adolescents with type 1 diabetes in chronic poor metabolic control: a randomized controlled trial. Diabetes Care. 2005 Jul;28(7):1604-10. doi: 10.2337/diacare.28.7.1604. PMID 15983308
- [Result] Ellis DA, Frey MA, Naar-King S, Templin T, Cunningham PB, Cakan N. The effects of multisystemic therapy on diabetes stress among adolescents with chronically poorly controlled type 1 diabetes: findings from a randomized, controlled trial. Pediatrics. 2005 Dec;116(6):e826-32. doi: 10.1542/peds.2005-0638. PMID 16322140
- [Result] Ellis DA, Naar-King S, Frey M, Templin T, Rowland M, Cakan N. Multisystemic treatment of poorly controlled type 1 diabetes: effects on medical resource utilization. J Pediatr Psychol. 2005 Dec;30(8):656-66. doi: 10.1093/jpepsy/jsi052. Epub 2005 Mar 3. PMID 16260435
- [Result] Naar-King S, Podolski CL, Ellis DA, Frey MA, Templin T. Social ecological model of illness management in high-risk youths with type 1 diabetes. J Consult Clin Psychol. 2006 Aug;74(4):785-9. doi: 10.1037/0022-006X.74.4.785. PMID 16881786
- [Result] Naar-King S, Idalski A, Ellis D, Frey M, Templin T, Cunningham PB, Cakan N. Gender differences in adherence and metabolic control in urban youth with poorly controlled type 1 diabetes: the mediating role of mental health symptoms. J Pediatr Psychol. 2006 Sep;31(8):793-802. doi: 10.1093/jpepsy/jsj090. Epub 2005 Dec 1. PMID 16322274
- [Result] Ellis DA, Templin T, Naar-King S, Frey MA, Cunningham PB, Podolski CL, Cakan N. Multisystemic therapy for adolescents with poorly controlled type I diabetes: Stability of treatment effects in a randomized controlled trial. J Consult Clin Psychol. 2007 Feb;75(1):168-74. doi: 10.1037/0022-006X.75.1.168. PMID 17295576
- [Result] Ellis DA, Yopp J, Templin T, Naar-King S, Frey MA, Cunningham PB, Idalski A, Niec LN. Family mediators and moderators of treatment outcomes among youths with poorly controlled type 1 diabetes: results from a randomized controlled trial. J Pediatr Psychol. 2007 Mar;32(2):194-205. doi: 10.1093/jpepsy/jsj116. Epub 2006 May 4. PMID 16675714
- [Result] Cakan N, Ellis DA, Templin T, Frey M, Naar-King S. The effects of weight status on treatment outcomes in a randomized clinical trial of multisystemic therapy for adolescents with type 1 diabetes and chronically poor metabolic control. Pediatr Diabetes. 2007 Aug;8(4):206-13. doi: 10.1111/j.1399-5448.2007.00273.x. PMID 17659062
- [Derived] Ellis D, Naar-King S, Templin T, Frey M, Cunningham P, Sheidow A, Cakan N, Idalski A. Multisystemic therapy for adolescents with poorly controlled type 1 diabetes: reduced diabetic ketoacidosis admissions and related costs over 24 months. Diabetes Care. 2008 Sep;31(9):1746-7. doi: 10.2337/dc07-2094. Epub 2008 Jun 19. PMID 18566340